CLINICAL TRIAL: NCT00830609
Title: Effect of High Dose vs. Standard Dose of Ribavirin in Patients With Chronic Hepatitis C, Genotype 3, High Viral Load Without Rapid Virological Response
Brief Title: High Dose Versus Standard Dose of Ribavirin in Patients With Chronic Hepatitis C, Genotype 3
Acronym: DARGEN-3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Conrado Fernandez (Other)
Responsible Party: Sponsor-Investigator, Dr. Conrado Fernandez, MD, Hospital Universitario Fundación Alcorcón
Organization: Hospital Universitario Fundación Alcorcón (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROCHE FARMA S.A.
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C; Genotype 3; High viral load
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin; epoetin beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Active Comparator): Patients in this arm will receive standard of care (Peginterferon alfa 2A 180 mcg/weeks SC plus ribavirin 800 mg/day for 24 weeks).
  Interventions: Drug: Peginterferon alfa 2 A; Drug: ribavirin
- B1 (Experimental): After a period of 4 weeks with peginterferon alfa 2 a 180 mcg/week plus RBV 1600 mg/day (Induction phase), these patients will be allocated according to negativity or positivity of RNA-HCV at week 4. If RNA-HCV negative, treatment with peginterferon alfa 2 a 180 mcg/week plus RBV 800 mg/day (SOC) will be continued over 20 additional weeks (Arm B1). Epo β (450 IU/kg/week) will be administered as required to maintain hemoglobin > 12g/dL.
  Interventions: Drug: Peginterferon alfa 2 A; Drug: Peginterferon alfa 2 A, ribavirin + Epo Beta; Drug: Peginterferon alfa 2; Drug: ribavirin
- B2 (Experimental): If RNA-HCV at week 4 remains positive after the induction phase, then peginterferon alfa 2 a 180 mcg/week plus RBV 1600 mg/day will be continued for 20 additional weeks (Arm B2). Epo β (450 IU/kg/week) will be administered as required to maintain hemoglobin > 12g/dL.
  Interventions: Drug: Peginterferon alfa 2 A; Drug: Peginterferon alfa 2 A, ribavirin + Epo Beta; Drug: ribavirin

INTERVENTIONS:
Drug: Peginterferon alfa 2 A — Peginterferon alfa 2 A 180 mcg/week SC plus Ribavirin 800 mg/day po (Control Group) Peginterferon alfa 2 A 180 mcg/week SC plus Ribavirin 1,600 mg/day po plus Epoetin β (450 IU/kg/week) SC over 4 weeks (Arm B1) Peginterferon alfa 2 A 180 mcg/week SC plus Ribavirin 1,600 mg/day po plus Epo beta 450 UI over four weeks (Arm B1) If RNA-HCV positive at week 4, Peginterferon alfa 2 A 180 mcg/week SC plus Ribavirin 1,600 mg/day plus Epo beta 450 UI to keep Hb>12 g/dL if required over 20 additional weeks (Arm B2)
  Other Names: Pegasys
Drug: Peginterferon alfa 2 A, ribavirin + Epo Beta — Ribavirin 1,600 mg/day plus peginterferon alfa 2A 180 mcg/week plus Epo beta 450 IU/Kg/day to maintain Hb>12g/dl over 4 or 24 weeks
  Other Names: Pegasys
  Arms: B1; B2
Drug: ribavirin — RBV 1600 mg/day 24 weeks
  Other Names: peginterferon alfa 2 a; Epoetin beta
  Arms: B2
Drug: ribavirin — ribavirin 800 mg/day for 24 weeks
  Other Names: Pegasys
  Arms: A
Drug: Peginterferon alfa 2 — Peginterferon alfa 2 a 180 mcg/week for 4 weeks and then peginterferon alfa 2A for 20 weeks
  Other Names: Pegasys
  Arms: B1
Drug: ribavirin — RBV 1600 mg/day 4 weeks and then ribavirin 800 mg/day 20 weeks
  Other Names: Pegasys
  Arms: B1

SUMMARY:
The rate of sustained virological response (SVR) in patients with chronic hepatitis C, genotype 3, high viral load and without rapid virological response (RNA-HCV negative at week 4) is low. Standard of care of these patients include treatment with weekly peginterferon plus 800 mg/day of ribavirin (RBV). Extended treatment to 48 weeks does not provide more clinical benefit than the standard duration. The main hypothesis is that higher dose of ribavirin may be better in terms of SVR than the standard dose.

DETAILED DESCRIPTION:
Aims:

1. Efficacy 1.1) Rate of RNA-HCV negative at week 4 and 24 in each arm. 1.2) Rate of SVR in each arm.
2. Safety 2.1) Rate of adverse effects in each arm.

Design: Randomized controlled trial.

Patients will be randomly allocated into three arms:

Arm A : Peginterferon α-2a (180 μg/week)SC. plus Ribavirin (800 mg/day) p.o. over 24 weeks.

Arm B: Peginterferon α-2a (180 μg/week) plus Ribavirin (1600 mg/day) with support of Epoetin β (450 IU/kg/week) SC over 4 weeks:

B1.- If RNA-HCV undetectable at week 4, standard of care will be continued (Peginterferon α-2a, 180 μg/wee plus Ribavirin (800 mg/day) over 20 additional weeks).

B2.- If RNA-HCV were detectable at week 4, treatment will be continued with peginterferon α-2a (180 μg/week) plus RBV(1,600 mg/day) plus Epoetin β (450 UI/kg/week) over 20 additional weeks.

Sample size: 111 patients. To increase the SVR from 50% to 75%. Beta: 0.1; alfa: 0.05; Loss: 15%.

Randomization will be 1:2, 37 patients in Group A and 74 patients in group B.

ELIGIBILITY:
Inclusion Criteria:

* HCV Genotype 3
* RNA-HCV > > 600.000 IU/ml.
* Compromise to use contraceptive measures on treatment until 6 months after the end of treatment.

Exclusion Criteria:

* Pregnant or breastfeeding females.
* Concurrent treatment with antineoplastic or immunomodulatory agents, including corticosteroids or radiation therapy over the last 6 months before starting the trial
* Treatment with investigational drugs < 6 weeks before starting the trial
* Chronic liver disease other than hepatitis C.
* Evidence of hepatocellular carcinoma.
* Evidence of carcinoma hepatocellular
* Decompensated liver disease
* Baseline Neutrophil count < 1500/cc; or Platelet count < 90,000/cc
* Baseline Hemoglobin <12 g/dL in females o <13 g/dL in males.
* Increased risk of anemia(Eg, thalassemia, spherocytosis..).
* Ischemic heart disease or cerebrovascular disease.
* Serum creatinine >1.5 times upper limit of normality.
* History of severe psychiatric conditions (Major antidepressives or neuroleptic drugs required for major depression or psychosis), suicide attempts or psychiatric disability .
* History of convulsive disorders.
* Immunological conditions.
* Chronic Obstructive Lung Disease with limited functionality
* Severe heart disease or congestive cardiac insufficiency cardiopathy grave.
* Advanced atherosclerosis
* Solid organ or bone marrow transplant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2008-11; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Rate of patients with RNA-HCV negative in each arm at week 24 after the end of treatment. | 1 year

SECONDARY OUTCOMES:
Rate of patients with undetectable RNA-HCV in each arm at week 4 and 24 of treatment. Rate of adverse effects in each arm. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Conrado M Fernandez-Rodriguez, Study Director — Hospital Universitario Fundacion Alcorcon; University Rey Juan Carlos.
Locations (28):
- Spain (28):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Barcelona
  - Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Parc Taulí, Sabadell, Barcelona
  - Hospital Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Reina Sofía, Córdoba, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - Hospital San Cecilio, Granada, Granada
  - Hospital de Donostia, Donostia / San Sebastian, Guipuzcoa
  - Hospital de León, León, León
  - Hospital Fundación Alcorcón, Alcorcón, Madrid
  - Hospital de Getafe, Getafe, Madrid
  - Hospital La Princesa, Madrid, Madrid
  - Hospital Gregorio Marañon, Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - Hospital Costa del Sol, Marbella, Málaga
  - Hospital Clínico Universitario Virgen de la Victoria, Málaga, Málaga
  - Hospital Central de Asturias, Oviedo, Oviedo
  - Hospital Clinico Universitario de Salamanca, Salamanca, Salamanca
  - Hospital de Valme, Seville, Sevilla
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid, Valladolid
  - Hospital Santiago Apóstol, Vitoria-Gasteiz, Vitoria
  - Hospital Clínico de Zaragoza, Zaragoza, Zaragoza
  - Hospital Miguel Servet, Zaragoza, Zaragoza

REFERENCES:
- [Derived] Fernandez-Rodriguez CM, Morillas RM, Masnou H, Navarro JM, Barcena R, Gonzalez JM, Martin-Martin L, Poyato A, Miquel-Planas M, Jorquera F, Casanovas T, Salmeron J, Calleja JL, Sola R, Alonso S, Planas R, Romero-Gomez M. Randomized clinical trial comparing high versus standard dose of ribavirin plus peginterferon alfa-2a in hepatitis C genotype 3 and high viral load. Dargen-3 study. Gastroenterol Hepatol. 2014 Jan;37(1):1-8. doi: 10.1016/j.gastrohep.2013.10.005. Epub 2013 Dec 17. PMID 24360571